CLINICAL TRIAL: NCT07402811
Title: Mindfulness-Based Intervention for Pain and Sleep in Adolescents and Young Adults With Sickle Cell Disease
Acronym: REMedy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Dahee Wi, Postdoctoral Research Associate, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY2024-0914-MOD007; K99NR021195-01A1 (NIH)
Record Dates: First submitted 2026-01-26; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain; Sickle Cell Disease; Sleep Disturbance
Keywords: sleep; mindfulness-based intervention; mobile health; feasibility study; pain management
MeSH Terms: conditions — Chronic Pain; Anemia, Sickle Cell; Parasomnias; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-based intervention (Experimental): Participants are assigned to a single study arm and receive a mindfulness-based mobile intervention delivered via a smartphone application over approximately 8 weeks.
  Interventions: Behavioral: Mobile bindfulness-based intervention

INTERVENTIONS:
Behavioral: Mobile bindfulness-based intervention — Participants receive a mindfulness-based mobile intervention designed to support symptom management related to pain and sleep. The intervention is delivered via a smartphone application and includes structured mindfulness content such as guided meditation and brief mindfulness exercises. Participants are asked to engage with the intervention over an approximately 8-week period. The study evaluates feasibility and acceptability.

SUMMARY:
This study examines the feasibility and acceptability of a mindfulness-based mobile intervention designed to support pain and sleep management among adolescents and young adults with sickle cell disease. Chronic pain and sleep problems are common in this population and can negatively affect daily functioning and quality of life. Participants will use a smartphone-based mindfulness program that includes structured modules and guided mindfulness exercises over an approximately 8-week period. The study aims to evaluate whether the intervention is feasible and acceptable for adolescents and young adults with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 15-39 years
* Have been diagnosed with SCD
* Are able to speak and understand English
* Are able to complete questionnaires with minimal or no assistance from a caregiver
* Report pain and/or sleep problems as assessed by the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) short forms
* Have access to the internet on a smartphone, tablet, or computer

Exclusion Criteria:

* Individuals who have significant cognitive limitations that will impair their ability to use and understand the MBI, as per their health care provider or caregiver
* Are currently receiving an MBI or have received more than 4 sessions of any MBI in the 6 months prior to the screening

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Participant retention rate | At 8 weeks (post-intervention)
  Percentage of enrolled participants who remain in the study through the 8-week intervention period
Attrition rate and reasons for withdrawal | Throughout the 8-week intervention period
  Percentage of participants who withdraw from the study and documented reasons for withdrawal
Weekly module completion rate | At 8 weeks (post-intervention)
  Percentage of assigned weekly modules completed by participants
Acceptability of the Mindfulness-Based Intervention | At 8 weeks (post-intervention)
  Acceptability of the digital mindfulness-based intervention assessed using a study-specific acceptability questionnaire. The questionnaire measures multiple dimensions including comfort level, effort required to engage, perceived fairness for patients with sickle cell disease, perceived effectiveness for pain and sleep management, clarity of intervention purpose, confidence in the intervention, interference with other priorities, and overall acceptability. The questionnaire uses 5-point rating scales for all items. The questionnaire also includes open-ended questions about device use, suggested improvements, and helpful and unhelpful aspects of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dahee Wi, PhD, RN, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No